CLINICAL TRIAL: NCT02724111
Title: Comparison of Operating Conditions, Postoperative Recovery and Overall Satisfaction Between Deep and Restricted Neuromuscular Blockade for Spinal Surgery Under General Anesthesia
Brief Title: Effect of Neuromuscular Blockade on Operating Conditions and Overall Satisfaction During Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Byung Gun Lim, Associate Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KUGH15297-002
Record Dates: First submitted 2016-03-24; First posted 2016-03-31 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Neuromuscular Blockade; Surgery; Anesthesia; Spinal Diseases
Keywords: Neuromuscular blockade; Surgical rating scale; Rocuronium; Sugammadex; Spinal surgery; General anesthesia
MeSH Terms: conditions — Spinal Diseases | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- deep neuromuscular blockade (Experimental): This arm will be given sufficient dose of rocuronium. In this Arm group, rocuronium will be administered to maintain deep neuromuscular blockade [NMB] (train-of-four [TOF] count 0, post-tetanic count [PTC] of 1-2 twitches) until the end of surgery and the reversal of NMB will be performed by sugammadex 4 mg/kg at the end of surgery'.
  Interventions: Drug: sufficient dose of rocuronium
- restricted neuromuscular blockade (Active Comparator): This arm will not be given sufficient dose of rocuronium. In this Arm group, sugammadex will be administered according to the prescribing indications (4 mg/kg for deep neuromuscular blockade [NMB] state or 2 mg/kg for moderate NMB or less) to reverse the NMB 10 min after position change (sugammadex 10 min after position change [a prone position]). Thereafter, muscle relaxants will not be injected any more throughout the surgery except the following situations: If the patients show any body movement during surgery or if surgeons express any complaint about muscle tone (the muscle tone: grade 3), rescue rocuronium 5 mg will be administered and the number of body movements and rescue rocuronium administration (dose) will be recorded.
  Interventions: Drug: sugammadex 10 min after position change

INTERVENTIONS:
Drug: sufficient dose of rocuronium
  Other Names: sugammadex at the end of surgery
  Arms: deep neuromuscular blockade
Drug: sugammadex 10 min after position change
  Other Names: restricted dose of rocuronium
  Arms: restricted neuromuscular blockade

SUMMARY:
The investigators aim to investigate operating conditions, postoperative recovery and overall satisfaction of surgeons between deep neuromuscular blockade (NMB) group and restricted NMB group during spinal surgery under general anesthesia. The investigators hypothesize that this study can present good surgical conditions, postoperative recovery outcomes and overall satisfaction of surgeons in deep NMB group, thereby proving the advantages of deep NMB as well as flaws of restricted NMB in spine surgeries.

DETAILED DESCRIPTION:
* Group treatment (Arms): group treated with restricted neuromuscular blockade (NMB) (Group RB); group treated with deep NMB (Group DB) → randomized allocation (subjects: motor-evoked potential [MEP] not monitored surgeries)
* Inclusion criteria: American Society of Anesthesiologists (ASA) physical status I-II adults, aged 18-75 years, scheduled for elective spinal surgery (cervical or lumbar surgeries which have lesions no more than 3 spinal levels and not monitored by MEP) of duration >1 hour and prone position under total intravenous anesthesia (TIVA).
* Exclusion criteria: Pregnancy, the receipt of medication known to interfere with neuromuscular blockade, diseases affecting neuromuscular transmission, and the history of hypersensitivity on rocuronium or sugammadex. The patients who will have hemodynamic instability, mean blood pressure increase or fall of > 30% from baseline (lasting for more than 5min), and blood loss > 1 L during surgery, and MEP monitored surgeries.
* Outcome Measures

  * Primary outcome: Mean value of peak inspiratory pressure recorded every 15 minutes.
  * Secondary outcomes:

    1. The number of body movements (including cough or any diaphragm movement).
    2. The degree of bleeding of each patient scaled by surgeons (Intraoperative scale for assessment of operating condition of surgical field: 0 - No bleeding, 1 - Slight bleeding - no suctioning of blood required, 2 - Slight bleeding - occasional suctioning required but not threatened the operative field, 3 - Slight-bleeding - frequent suctioning of blood was required that threatens the operative field a few seconds after suctioning, 4 - Moderate bleeding - frequent suctioning of blood was required which threatens the operative field directly after suctioning, 5 - Sever bleeding - continuous suctioning of blood was required which severely threatened the operative field make the surgery not possible).
    3. The muscle tone of each patient scaled by surgeons (1: muscle tone is good, suitable for surgery; 2: muscle tone is moderate, but do not affect the operation; 3: muscle tone is hard, making the operation difficult.).

       * Three time-points of assessment of the muscle tone: ① At the placement of back muscle retractor for opening the operating site after the skin and subcutaneous incision, ② At the screw insertion through the pedicle of spine during surgery, ③ At the other period (overall muscle tone).
    4. Mean value of pressure of back muscle retractor placed in the operating site (recorded every 15 minutes): measured by the pressure probe placed between the retractor and the back muscle.
    5. Overall satisfaction of surgeons for the surgical condition will be assessed by the surgeons who perform surgery using numerical rating scale (NRS; 1-10) after surgery.
    6. Recovery profiles including eye opening time, extubation time and sedation score (the Observer's Assessment of Alertness/ Sedation (OAA/S) score; awake, 5 to unresponsive, 1) every 10 min for 1 hour at postanesthesia care unit (PACU).
    7. Postoperative adverse events

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II adult patients scheduled for elective spinal (cervical or lumbar) surgery under general anesthesia

Exclusion Criteria:

* Pregnancy
* Present medication known to interfere with neuromuscular blockade
* Diseases affecting neuromuscular transmission
* History of hypersensitivity on rocuronium or sugammadex
* Emergent spinal surgery
* Spinal surgeries which have lesions more than 3 spinal levels
* Spinal surgeries which have duration less than 1 hour
* Spinal surgeries which are not performed under prone position
* Spinal surgeries which are not performed under total intravenous anesthesia (TIVA).
* Patients who will have hemodynamic instability (mean blood pressure increase or fall of > 30% from baseline lasting for more than 5 min) during surgery
* Patients who will have blood loss > 1 L during surgery
* MEP monitored spinal surgeries

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byung Gun Lim, Ph.D., Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a single-site study recruited and performed at Korea University Guro Hospital, a general hospital, Seoul, South Korea, from 15 May 2016 to 16 February 2017.
Pre-assignment Details: No enrolled participants were excluded from the study before assignment to arms or groups.
Groups:
- Deep Neuromuscular Blockade: This arm will be given sufficient dose of rocuronium. In this Arm group, rocuronium will be administered to maintain deep neuromuscular blockade [NMB] (train-of-four [TOF] count 0, post-tetanic count [PTC] of 1-2 twitches) until the end of surgery and the reversal of NMB will be performed by sugammadex 4 mg/kg at the end of surgery'.
  sufficient dose of rocuronium
- Restricted Neuromuscular Blockade: This arm will be given restricted (not sufficient) dose of rocuronium. In this Arm group, sugammadex will be administered according to the prescribing indications (4 mg/kg for deep neuromuscular blockade [NMB] state or 2 mg/kg for moderate NMB or less) to reverse the NMB 10 min after position change (sugammadex 10 min after position change [a prone position]). Thereafter, muscle relaxants will not be injected any more throughout the surgery except the following situations: If the patients show any body movement during surgery or if surgeons express any complaint about muscle tone (the muscle tone: grade 3), rescue rocuronium 5 mg will be administered and the number of body movements and rescue rocuronium administration (dose) will be recorded.
  sugammadex 10 min after position change
Period: Overall Study
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade
Started | 45 | 45
Completed | 43 | 40
Not Completed | 2 | 5
Not completed — Protocol Violation | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Deep Neuromuscular Blockade: This arm will be given sufficient dose of rocuronium. In this Arm group, rocuronium will be administered to maintain deep neuromuscular blockade [NMB] (TOF count 0, post-tetanic count [PTC] of 1-2 twitches) until the end of surgery and the reversal of NMB will be performed by sugammadex 4 mg/kg at the end of surgery'.
  sufficient dose of rocuronium
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade | Total
Number analyzed (Participants) | 43 | 40 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 31 | 61
  >=65 years | 13 | 9 | 22
Age, Continuous [Median (Full Range); unit: years] | 61 [37 to 75] | 60 [30 to 75] | 60 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 43 | 40 | 83
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 43 | 40 | 83
Height (m) [Mean (Standard Deviation); unit: meter] | 1.59 (0.07) | 1.58 (0.08) | 1.59 (0.07)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 59.8 (8.5) | 60 (6.9) | 59.9 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Mean Value of Peak Inspiratory Pressure
Description: This outcome is the mean value of the peak inspiratory pressure measured at each 15 minute during the anesthesia, which can reflect the degree of the tone of respiratory muscles. As muscle tone increases, airway pressure usually increases due to increased tone of abdominal muscle and respiratory muscles including diaphragm. The longer the surgery goes, the higher the airway pressure gets. Also, as neurospinal surgeries are operated in the prone position, the potential for increased airway pressure is high. As airway pressure gets higher, intrathoracic pressure and intraabdominal pressure also become higher. These consequences may bring about similar results with detrimental effects derived from marked increase in intraabdominal pressure in laparoscopic abdominal surgeries
Time Frame: Every 15 minutes during anesthesia, up to 3 hours
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade
Number analyzed (Participants) | 43 | 40
cmH2O | 18.4 (1.1) | 20.2 (1.1)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade vs Restricted Neuromuscular Blockade; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Mean Value of Pressure of Back Muscle Retractor
Description: Mean value of pressure of back muscle retractor placed in the operating site (recorded every 15 minutes during the placement of the retractor): measured by the pressure probe placed between the retractor and the back muscle.
Time Frame: Every 15 minutes at the period of the retractor placement during surgery, up to 2 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade
Number analyzed (Participants) | 43 | 40
mmHg | 81.2 (9.1) | 100 (7.3)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade vs Restricted Neuromuscular Blockade; Test type: Superiority; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Overall Satisfaction of Surgeons for the Surgical Condition
Description: Overall satisfaction of surgeons for the surgical condition will be assessed by the surgeons who perform surgery using numerical rating scale (NRS; 1-10) after surgery (1, worst; 10, best).
Time Frame: After surgery
Measure: Mean (Standard Deviation); unit: Scores on a scale (NRS; 1-10)
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade
Number analyzed (Participants) | 43 | 40
Scores on a scale (NRS; 1-10) | 8 (1.3) | 3.1 (1.2)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade vs Restricted Neuromuscular Blockade; Test type: Superiority; p < 0.001, t-test, 2 sided

4. Secondary Outcome: The Muscle Tone
Description: The muscle tone of each patient at the screw insertion through the pedicle of spine during surgery scaled by surgeons (1: muscle tone is good, suitable for surgery; 2: muscle tone is moderate, but do not affect the operation; 3: muscle tone is hard, making the operation difficult.).
Time Frame: at the screw insertion through the pedicle of spine during surgery
Measure: Mean (Standard Deviation); unit: Scores on a scale (NRS; 1-3)
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade
Number analyzed (Participants) | 43 | 40
Scores on a scale (NRS; 1-3) | 1.3 (0.7) | 2.5 (0.7)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade vs Restricted Neuromuscular Blockade; Test type: Superiority; p < 0.001, Chi-squared

5. Secondary Outcome: The Number of Body Movements
Description: The number of body movements (including cough or any diaphragm movement) observed during the surgery.
Time Frame: At the occurrence of the event during surgery, up to 3 hours
Measure: Mean (Standard Deviation); unit: number of event
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade
Number analyzed (Participants) | 43 | 40
number of event | 0 (0) | 2 (1)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade vs Restricted Neuromuscular Blockade; Test type: Superiority; p < 0.001, Chi-squared

6. Secondary Outcome: The Degree of Bleeding
Description: 2.The degree of bleeding of each patient scaled by surgeons (Intraoperative scale for assessment of operating condition of surgical field: 0 - No bleeding, 1 - Slight bleeding - no suctioning of blood required, 2 - Slight bleeding - occasional suctioning required but not threatened the operative field, 3 - Slight-bleeding - frequent suctioning of blood was required that threatens the operative field a few seconds after suctioning, 4 - Moderate bleeding - frequent suctioning of blood was required which threatens the operative field directly after suctioning, 5 - Severe bleeding - continuous suctioning of blood was required which severely threatened the operative field make the surgery not possible).
Time Frame: Continuously observed during the whole period of surgery, up to 3 hours
Measure: Mean (Standard Deviation); unit: Scores on a scale (NRS; 0-5)
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade
Number analyzed (Participants) | 43 | 40
Scores on a scale (NRS; 0-5) | 1.8 (0.7) | 3.3 (0.7)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade vs Restricted Neuromuscular Blockade; Test type: Superiority; p < 0.001, t-test, 2 sided

7. Secondary Outcome: Recovery Time (Time to Reach Sedation Score 5 at Postanesthesia Care Unit (PACU).
Description: the time to reach sedation score 5 (the Observer's Assessment of Alertness/ Sedation (OAA/S) score; awake, 5 to unresponsive, 1) at PACU
Time Frame: every 10 min for 1 hour at PACU.
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade
Number analyzed (Participants) | 43 | 40
minute | 10.5 (7.9) | 17 (11.4)
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade vs Restricted Neuromuscular Blockade; Test type: Superiority; p = 0.06, t-test, 2 sided

8. Secondary Outcome: Adverse Events : The Postoperative Nausea and Vomiting Occurrence in Subject
Description: The occurrence of any adverse events was recorded in the post-anesthesia care unit (PACU) and a ward during the postoperative 24 hours.
Time Frame: during the postoperative 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade
Number analyzed (Participants) | 43 | 40
Participants | 11 | 8
Statistical Analysis 1: Comparison: Deep Neuromuscular Blockade vs Restricted Neuromuscular Blockade; Test type: Superiority; p = 0.202, Chi-squared

ADVERSE EVENTS:
Time Frame: during the postoperative 24 hours
Description: Same.
Arm/Group | Deep Neuromuscular Blockade | Restricted Neuromuscular Blockade
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/40
Other Adverse Events (participants affected / at risk) | 11/43 | 8/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deep Neuromuscular Blockade (N=43) | Restricted Neuromuscular Blockade (N=40)
nausea or vomiting (Gastrointestinal disorders) | 11 | 8 — This adverse event is the postoperative nausea and vomiting occurred during the postoperative 24 hours. The symptoms were all resolved well after administration of antiemetics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT02724111/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT02724111/SAP_001.pdf
  • Informed Consent Form (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT02724111/ICF_002.pdf